CLINICAL TRIAL: NCT00369005
Title: Randomized Trial of Liberal Versus Restrictive Guidelines for Red Blood Cell Transfusion in Preterm Infants
Brief Title: Liberal Versus Restrictive Transfusion Guidelines for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IowaBell001; P01HL046925 (NIH); M01RR000059 (NIH)
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Infant, Premature; Anemia; Intracranial Hemorrhages; Leukomalacia, Periventricular; Apnea
Keywords: Transfusions; Erythrocyte; Anemia; Brain; Infant, Premature
MeSH Terms: conditions — Premature Birth; Anemia; Intracranial Hemorrhages; Leukomalacia, Periventricular; Apnea

INTERVENTIONS:
Procedure: Red blood cell transfusion guidelines

SUMMARY:
The purpose of this study was to determine whether restrictive guidelines for red blood cell (RBC) transfusions for preterm infants can reduce the number of transfusions without adverse consequences.

DETAILED DESCRIPTION:
Design, Setting, and Patients. We enrolled 100 hospitalized preterm infants with birth weights 500 to 1300 g into a randomized clinical trial comparing two levels of hematocrit threshold for RBC transfusion.

Intervention. The infants were randomly assigned to either the liberal or the restrictive transfusion group. For each group, transfusions were given only when the hematocrit fell below the assigned value. In each group, the transfusion thresholds decreased with improving clinical status.

Main Outcome Measures. We recorded the number of transfusions, the number of donor exposures, and various clinical and physiological outcomes.

Results. Infants in the liberally transfused group received more RBC transfusions, mean 5.2 (SD 4.5) vs 3.3 (SD 2.9) in the restrictive transfusion group (P=0.025). However, the number of donors to whom the infants were exposed was not significantly different, mean 2.8 (SD 2.5) vs 2.2 (SD 2.0). There was no difference between the groups in the percentage of infants who avoided transfusions altogether, 12% in the liberal transfusion group vs 10% in the restrictive group. Infants in the restrictive group were more likely to have intraparenchymal brain hemorrhage or periventricular leukomalacia (P=0.012), and they had more frequent episodes of apnea (P=0.004), including both mild and severe episodes.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant
* Birth weight 500-1300 grams

Exclusion Criteria:

* Alloimmune hemolytic disease
* Congenital heart disease
* Other major birth defect requiring surgery
* Chromosomal abnormality
* Thought to be facing imminent death
* Parental philosophical or religious objections to transfusion
* More than 2 transfusions before enrollment
* Participation in other research study with potential impact on this study

Ages: 0 Years to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 1992-12; Study Completion 1999-06

PRIMARY OUTCOMES:
number of red blood cell transfusions
number of transfusion donors

SECONDARY OUTCOMES:
survival to discharge
patent ductus arteriosus
germinal matrix or intraventricular hemorrhage
periventricular leukomalacia
retinopathy of prematurity
bronchopulmonary dysplasia
duration of assisted ventilation
duration of supplemental oxygen therapy
number and frequency of all apnea episodes
number and frequency of apnea episodes requiring tactile stimulation
number and frequency of apnea episodes requiring assisted ventilation
number and frequency of apnea episodes during the 24 hours before and after each transfusion
time to regain birth weight
time to double birth weight
length of hospitalization
hemoglobin
hematocrit
reticulocyte count
oxygen saturation (pulse oximetry)
cardiac output (echocardiography)
blood lactic acid
plasma erythropoietin
serum ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. Bell, M.D., Principal Investigator — University of Iowa

REFERENCES:
- [Result] Bell EF, Strauss RG, Widness JA, Mahoney LT, Mock DM, Seward VJ, Cress GA, Johnson KJ, Kromer IJ, Zimmerman MB. Randomized trial of liberal versus restrictive guidelines for red blood cell transfusion in preterm infants. Pediatrics. 2005 Jun;115(6):1685-91. doi: 10.1542/peds.2004-1884. PMID 15930233
- [Derived] Nopoulos PC, Conrad AL, Bell EF, Strauss RG, Widness JA, Magnotta VA, Zimmerman MB, Georgieff MK, Lindgren SD, Richman LC. Long-term outcome of brain structure in premature infants: effects of liberal vs restricted red blood cell transfusions. Arch Pediatr Adolesc Med. 2011 May;165(5):443-50. doi: 10.1001/archpediatrics.2010.269. Epub 2011 Jan 3. PMID 21199970